CLINICAL TRIAL: NCT01137838
Title: Changes in the Use of Opioids, Antidepressants, and Benzodiazepines in Rheumatoid Arthritis Patients Treated With Biologic Agents
Status: Completed | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Study Director, Bristol-Myers Squibb
Other Study IDs: IM101-238
Record Dates: First submitted 2010-06-02; First posted 2010-06-07 (Estimated); Last update posted 2011-05-17 (Estimated); Status verified 2011-05

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Patients with RA and new to abatacept
- Patients with RA and new to infliximab
- Patients with RA and new to etanercept
- Patients with RA and new to adalimumab

SUMMARY:
To compare the proportion of rheumatoid arthritis (RA) patients prescribed opioids, benzodiazepines, and antidepressants before versus after starting each of the following biologics: abatacept, infliximab, etanercept, adalimumab, utilizing an administrative claims database.

ELIGIBILITY:
Inclusion Criteria:

* ICD 9 diagnosis RA 714.0
* Documented first biologic prescription ("index" prescription) for abatacept, infliximab, etanercept, or adalimumab
* Continuous therapy (gap between scripts no greater than 150% days supply) for minimum 6 months from index
* Prescription claims data available for 6 months before and 12 months after index biologic prescription
* Continuous eligibility for 6 months before and 12 months after index biologic prescription

Exclusion Criteria:

* Prescription claims for another biologic during the observation period (including rituximab and anakinra)
* Prescriptions not continuous for at least 6 months

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Commercial insurance claims database
Sampling Method: Non-Probability Sample
Enrollment: 1810 (Actual)
Dates: Start 2009-10; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Proportion of RA patients prescribed opioids, benzodiazepines, and antidepressants | 0-6 months after index biologic prescription
Proportion of RA patients prescribed opioids, benzodiazepines, and antidepressants | 7-12 months after index biologic prescription

SECONDARY OUTCOMES:
Prevalence of depression and/or anxiety (ICD-9 diagnosis code) | Between 0-6 months after index biologic prescription
Prevalence of depression and/or anxiety (ICD-9 diagnosis code) | 7-12 months after index biologic prescription

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb

REFERENCES:
- See also: BMS Clinical Trials Disclosure — http://www.bms.com/clinical_trials/Pages/home.aspx
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx
- See also: For FDA Safety Alerts and Recalls refer to the following link: http://www.fda.gov/MEDWATCH/safety.htm — http://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm